CLINICAL TRIAL: NCT01020682
Title: Apathy in Parkinson Disease: Clinical, Physiopathological and Pharmacological Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Délégation à la recherche clinique, CHU de grenoble
Other Study IDs: APATHIE
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Apathy in Parkinson Disease
Keywords: apathy; parkinson; agonist dopaminergic
MeSH Terms: conditions — Lethargy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Apathy has been reported to occur after subthalamic nucleus stimulation (STN-DBS), a treatment of motor complications in advanced Parkinson's disease (PD). It is not known whether postoperative apathy is related to dopamine withdrawal or a side effect of STN DBS. The researchers investigated potential predictors of apathy, and the effect of dopamine agonist treatment.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease

Exclusion Criteria:

* Mattis scale < 130
* Beck scale > 20

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2005-01; Primary Completion 2006-02 (Actual); Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital neurologique, Lyon, France